CLINICAL TRIAL: NCT04102553
Title: Phase III Study of F-18-PSMA-1007 vs F-18-Fluorocholine PET to Compare the Detection Rate of Prostate Cancer Lesions in Patients With Biochemical Recurrence After Previous Definitive Treatment for Localized Prostate Cancer
Brief Title: F-18-PSMA-1007 Versus F-18-Fluorocholine PET in Patients With Biochemical Recurrence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ABX advanced biochemical compounds GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: ABX-CT-301
Record Dates: First submitted 2019-09-24; First posted 2019-09-25 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Prostate Cancer; Prostate Cancer Recurrent
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F-18-PSMA-1007 (Experimental): Patients will receive F-18-PSMA-1007 PET/CT first, followed by F-18-Fluorocholine PET/CT.
  Interventions: Drug: F-18-PSMA-1007; Drug: F-18-Fluorocholine
- F-18-Fluorocholine (Active Comparator): Patients will receive F-18-Fluorocholine PET/CT first, followed by F-18-PSMA-1007 PET/CT.
  Interventions: Drug: F-18-PSMA-1007; Drug: F-18-Fluorocholine

INTERVENTIONS:
Drug: F-18-PSMA-1007 — Patients will receive F-18-PSMA-1007 PET/CT and F-18-Fluorocholine PET/CT in randomized order.
Drug: F-18-Fluorocholine — Patients will receive F-18-PSMA-1007 PET/CT and F-18-Fluorocholine PET/CT in randomized order.

SUMMARY:
This study evaluates the diagnostic performance and safety of F-18-PSMA-1007 and F-18-Fluorocholine PET/CT imaging in patients with suspected recurrence of prostate cancer after previous definitive treatment.

ELIGIBILITY:
Inclusion Criteria:

* male with original diagnosis of prostate carcinoma with prior definitive therapy
* suspicion of recurrence (3 consecutive PSA rises and/or PSA rise by 2.0 ng/mL or more above nadir after radiotherapy or cryotherapy and/or PSA rise by greater than 0.2 ng/mL after prostatectomy)
* life expectancy of 6 months or more as judged by the investigator
* willing and able to undergo all study procedures
* informed consent in writing (dated and signed)

Exclusion Criteria:

* age: less than18 years
* contraindications for F-18-Fluorocholine
* contraindications for any of the ingredients of F-18-PSMA-1007
* close affiliation with the investigational site; e.g. first-degree relative of the investigator
* at the time of enrolment into this study, participating in another therapeutic clinical trial or has completed study participation in another therapeutic clinical trial within 5 days of enrolment into this trial
* having been previously enrolled in this clinical trial
* mental conditions rendering the subject incapable to understand the nature, scope, and consequences of the trial
* being clinically unstable or requiring emergency treatment
* being considered a vulnerable person

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
To compare detection rate of metastatic prostate cancer lesions of F-18-PSMA-1007 versus F-18-Fluorocholine | Within 6 months after PET/CT

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Centre Jean Perrin Clermont-Ferrand, Clermont-Ferrand
  - Centre Léon Bérard LUMEN, Lyon
  - Hôpitaux de Brabois (Vandoeuvre-les-Nancy), Nancy
  - Hôpital Européen Georges-Pompidou, Paris
  - Hôpital Tenon, Paris
  - Hospices Civils de Lyon, Pierre-Bénite

REFERENCES:
- [Derived] Olivier P, Giraudet AL, Skanjeti A, Merlin C, Weinmann P, Rudolph I, Hoepping A, Gauthe M. Phase III Study of 18F-PSMA-1007 Versus 18F-Fluorocholine PET/CT for Localization of Prostate Cancer Biochemical Recurrence: A Prospective, Randomized, Crossover Multicenter Study. J Nucl Med. 2023 Apr;64(4):579-585. doi: 10.2967/jnumed.122.264743. Epub 2022 Nov 23. PMID 36418170